CLINICAL TRIAL: NCT05166252
Title: Are Offline Meals Healthy Meals? A Field Experiment to Promote Healthier Eating in Families
Acronym: OfflineMeals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Wuppertal (Other)
Collaborators: Max Planck Institute for Human Development (Other); University of Mannheim (Other)
Responsible Party: Principal Investigator, Theda Radtke, Prof. Dr., University of Wuppertal
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 180831
Record Dates: First submitted 2021-12-20; First posted 2021-12-21 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Health Behavior; Smartphone Addiction; Healthy Nutrition
MeSH Terms: conditions — Health Behavior; Internet Addiction Disorder

STUDY DESIGN:
Intervention Model Description: The study has an AB/BA crossover design, in which each participant receives the intervention and the control in a randomized order.
Who Masked: Participant
Masking Description: Families are assigned to the 2 conditions in a random order without knowing the aim of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 1. Installation of the study app.
  2. At the beginning of the meal, participants press a button within the App to start a time out from the smartphone at the beginning of a meal (i.e. calls and message are blocked and participants need to press an extra button in order to leave the app). The app instructs all other family members to turn off their phones and to put them away. Then, the participants are instructed to take a picture with their smartphone from the meal table.
  3. A time out from the smartphone starts, meaning that all functions of the phone are locked. The time-out is over as soon as the participant presses the "stop" button.
  4. A short questionnaire about the meal is sent via App to the participating family member when the smartphone is used again.
  5. During the whole period of the study the App tracks the smartphone behavior (i.e., frequency and duration of smartphone use and the specific applications used). Active comparator: control group
  Interventions: Behavioral: Time out from smartphone use during meal time
- Control group (Active Comparator): Control points in time include all parts as in the experimental group except for number 3.
  Interventions: Behavioral: Control condition

INTERVENTIONS:
Behavioral: Time out from smartphone use during meal time — One parent will be instructed to install a study app. Further, he/she press a button within the App to start a time out from the smartphone at the beginning of a meal (i.e. calls and message are blocked and the parent needs to press an extra button in order to leave the app). The app instructs all other family members to turn off their phones and to put them away. Then, the parent is instructed to take a picture with their smartphone from the "smartphone-free family meal table" . The time-out is over as soon as the parent presses the "stop" button.
  Arms: Experimental group
Behavioral: Control condition — The same as the experimental condition but without a timeout from smartphone use.
  Arms: Control group

SUMMARY:
First research findings suggest that the influence of digital media on children's and adolescents' health depends primarily on proper use and regulation. In line with Social Cognitive Theory, parents' own mobile device use is very important to regulate children's media use because parents are their children's role models. However, parents do not always behave as optimal role models: They use smartphones on playgrounds, in restaurants, as well as during family mealtimes. This usage of mobile devices leads to interruptions during face-to-face conversations or routines which is defined as "technoference". Studies among children and parents suggest that parental mobile device use is associated with fewer parent-child interactions. In addition, first studies investigated mobile device use at the dining table and showed that mothers had less interactions with their children during meal times when they used a mobile device compared to mothers who did not and their children were also less likely to try new and unfamiliar food. Along the same lines, lower parental mobile device use during mealtime is also associated with healthier body weight in children. AIM: Examination of the effect of a time out from smartphone use during a family meal on the parent-child interaction at the meal table and eating quality in comparison to family meals where participants use the smartphone as usual. DESIGN: The study is a within-family field experiment with daily assessments over 14 days (7 days for the experimental condition, 7 days for the control condition). Families will go through both, intervention and control condition with a break of 21 days in between. The assessment of the main and secondary outcomes is conducted at the baseline, over a 14 day daily diary phase and at the follow-up (directly after the daily diary phase). The sample will consist of 120 families with at least one child between the age of 6 to 14 years old. Only the participating adult in the study fills in the questionnaires. OUTCOMES: (Un)healthy eating and parent-child interaction constitute the main outcome, whereas technoference, mealtime duration, atmosphere at the meal table, and smartphone use frequency are secondary outcomes.

DETAILED DESCRIPTION:
Emerging mobile and digital technologies such as smartphones, tablets, wearables, and other mobile devices are an integral part in the daily lives of children, adolescents, and their families. The intensive use of mobile devices has both, positive aspects and negative side effects: The main advantages include access to information and making it easy to maintain social relationships. Potentially harmful risks for children include delays in small children's speech development, concentration disorders in primary school aged children or an increased consumption of sweet drinks and sweets. Especially parental media supervision is needed to regulate children's media use. In line with Social Cognitive Theory, parents' own mobile device use is also very important to regulate children's media use because parents are their children's role models. However, parents do not always behave as optimal role models: They use smartphones on playgrounds, as well as during family mealtimes. This usage of mobile devices leads to interruptions during face-to-face conversations or routines which is defined as "technoference". Studies among children and parents suggest that parental mobile device use is associated with fewer parent-child interactions. Especially using smartphones during shared meals could negatively influence interactions at the dining table as well as healthy eating habits in children. First findings suggest that the use of smartphones during family meals has detrimental effects on the family meal itself (e.g., interactions) as well as the health of the family members (e.g., diet quality and body weight). Importantly, these studies are all observational or cross-sectional, thus, experimental research is needed to understand whether taking the smartphone away from the family meal will actually lead to better interactions and healthier meals. While some experts suggest to ban smartphones from the dinner table, no one has systematically tested the effects. Thus, the aim of the proposed study is to experimentally test the effects of using smartphones at family meals versus banning them from the meal table and to examine potential mechanisms underlying this relation.

ELIGIBILITY:
Inclusion Criteria:

* One parent who 1. lives in a household with at least one child aged between 6 and 14 years 2. eats a family meal (shared meal) with this child at least 5 days/week 3. owns an Android smartphone 4. has mobile internet on the smartphone 5. uses the smartphone on a daily basis 6. uses the smartphone at least sometimes during shared meals 5. agrees on participating in the study.

Exclusion Criteria:

1. Insufficient knowledge of German of the participating family member
2. Involvement of the participating family member and/or child in a dietary program to reduce weight or plan to do so for the duration of the study.
3. Holidays during the intervention period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
(Un)healthy eating | Baseline, Daily Diaries (after Baseline assessment; 14 days in total), Follow up (35 days after the first daily diary assessment)
  Self-reported (un)healthy eating measured via intake of portions of fruits and vegetables, desserts, and sugar-sweetened beverages per day per child. Items according to Flückiger, L., Lieb, R., Meyer, A. H., Witthauer, C., & Mata, J. (2017). Day-to-day variations in health behaviors and daily functioning: Two intensive longitudinal studies. Journal of Behavioral Medicine, 40, 307-319.
Parent-child interaction | Daily Diaries (after Baseline assessment; 14 days in total)
  Parent-child interaction. Items according to: Mata, J., Dallacker, M., & Hertwig, R. (2018). A matter of time: Longer meal duration increases healthy eating in children. An experimental study. Invited presentation, conference of the German Society for Psychology, Frankfurt/ Main, Germany.

SECONDARY OUTCOMES:
Smartphone use | During the daily Diaries (after Baseline assessment; 14 days in total)
  Objective measurement: An app tracks general smartphone use (duration, frequency of unlocking, which applications were used)
Media use | Baseline, During the daily Diaries (after Baseline assessment; 14 days in total)
  Media use during meal time is measured with items from Knobl, V., Dallacker, M., Hertwig, R., & Mata, J. (manuscript submitted for publication). Happy and healthy: How family mealtime routines relate to child nutritional health.
Meal duration | Baseline, During the daily Diaries (after Baseline assessment; 14 days in total)
  Meal duration is measured with one item according to Knobl, V., Dallacker, M., Hertwig, R., & Mata, J. (manuscript submitted for publication). Happy and healthy: How family mealtime routines relate to child nutritional health.
Technoference | Baseline, Daily Diaries (after Baseline assessment; 14 days in total), Follow up (35 days after the first daily diary assessment)
  Technoference is measured according to McDaniel, B. T., & Coyne, S. M. (2016). "Technoference": The interference of technology in couple relationships and implications for women's personal and relational well-being. Psychology of Popular Media Culture, 5, 85-98. doi: 10.1037/ppm0000065
Child's distraction | Baseline, Daily Diaries (after Baseline assessment; 14 days in total), Follow up (35 days after the first daily diary assessment)
  Child's distraction is measured according to McDaniel, B. T., & Coyne, S. M. (2016). "Technoference": The interference of technology in couple relationships and implications for women's personal and relational well-being. Psychology of Popular Media Culture, 5, 85-98. doi: 10.1037/ppm0000065

CONTACTS AND LOCATIONS:
Overall Officials: Jutta Mata, Prof. Dr., Principal Investigator — University of Mannheim; Mattea Dallacker, Dr., Principal Investigator — Max Planck Institute for Human Development, Center for Adaptive Rationality; Theda Radtke, Prof. Dr., Principal Investigator — Uniersity of Wuppertal
Locations (1):
- Forsa, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No
We plan to provide the anonymized data set and the coding scheme.